CLINICAL TRIAL: NCT03942536
Title: The MOMENTUM Study (Monitoring Maternal Emergency Navigation and Triage on Mfangano) : A 12-month Community-based Cohort Study to Evaluate Delays in Access to Maternal and Newborn Emergency Care in Western Kenya
Brief Title: The MOMENTUM Study (Monitoring Maternal Emergency Navigation and Triage on Mfangano
Acronym: MOMENTUM
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Maseno University (Other)
Responsible Party: Sponsor
Other Study IDs: FMCH-2018-27289
Record Dates: First submitted 2019-01-14; First posted 2019-05-08 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Pregnancy; Neonatal Care; Emergency Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MNH Emergency Cohort: Participants will be either patients who have experienced a critical pregnancy-related, obstetric, or neonatal health emergency.
  Interventions: Other: Focus Group Discussion
- Birth Planning cohort: Pregnant women who complete an initial Birth Plan through the HN program within Mfangano Island East and South Sub-locations.
  Interventions: Other: Focus Group Discussion

INTERVENTIONS:
Other: Focus Group Discussion — At 12-month follow-up, a purposeful, convenience sample of study participants and their significant others, Community Health Workers trained as Health Navigators, and local program staff, will be invited by research staff to participate in focus group discussions to collect qualitative data on pregnancy care, experience of navigating obstetrical emergencies, financial hardships, and Health Navigation program feasibility/acceptability. Particular attention will be paid to recruiting study subjects involved in complex obstetrical emergencies, cases that involved significant delays in transfer of care, cases resulting in significant morbidity/mortality, as well as cases that involved efficient/successful care coordination, referral, and transportation.

SUMMARY:
This is an observational cohort study that will assess barriers influencing access to emergency pregnancy, obstetrical and neonatal care.

DETAILED DESCRIPTION:
Through a 12-month mixed methods, observational cohort study, investigators from Maseno University, University of Minnesota (UMN) and OHR-EKC will assess barriers influencing access to emergency pregnancy, obstetrical and neonatal care among patients seeking care at 9 health centers on Mfangano Island, as well as the preliminary impact and feasibility/acceptability of the HN approach for improving access to MNH services and shortening delays in care.

ELIGIBILITY:
Overall Inclusion Criteria:

* Must be ≥18 years of age as of the date of study eligibility, or qualify as an emancipated minor (ie: person aged less than 18 years who was married, pregnant, or a parent, consistent with Government of Kenya guidelines and previous research such as Kenya AIDS Indicator Survey-KAIS)
* Must be conversant with one of the commonly spoken languages within the study area (i.e. DhoLuo, Swahili or English; prior experience indicates that this represents >99% of the adult population)
* Must be willing to share confidential information about prenatal history, pregnancy course, obstetrical complications, clinical course, and experiences navigating health care system.
* Must have the ability to provide informed consent.

Emergency Cohort-Specific Criteria:

- Participants will be either patients who have experienced a critical pregnancy-related, obstetric, or neonatal health emergency, or appropriate family member in the case that patient is not able to participate in interview due to death or illness or other circumstance.

Birth Planning Cohort-Specific Criteria:

- All pregnant women who register a birth plan through the Health Navigation Birth Planning service will be eligible to enroll in the Birth Planning Cohort

Focus Group Cohort-Specific Criteria:

- All participants from the emergency cohort and the birth planning cohort will be eligible, as well as CHW volunteers, and OHR-EKC and MoH health facility staff

Exclusion Criteria:

* Individuals under the age of 18 and who do not qualify as emancipated minors
* Individuals who do not speak either English, Dholuo or Swahili
* Individuals who are not comfortable sharing confidential information about prenatal history, pregnancy course, obstetrical complications, clinical course, and experiences navigating health care system.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Research subjects must be pregnant
Study Population: Pregnant women, and CHW volunteers OHR-EKC and MoH health facility staff
Sampling Method: Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Assess time interval delays in access to emergency care among women and newborns who experience a critical health emergency | From subject enrollment through study completion, an average of 12 months.
  Quantify interval time delays in accessing emergency MNH care among women and newborns who experience a critical pregnancy-related, obstetrical, or neonatal health emergency on Mfangano Island Division.

CONTACTS AND LOCATIONS:
Overall Officials: Chas Salmen, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No